CLINICAL TRIAL: NCT06986278
Title: Transcranial Direct Current Stimulation Combined With Treadmill Training With Partial Body Weight Support in Patients With Multiple Sclerosis
Brief Title: tdCS Combined With Treadmill Training in Patients With Multiple Sclerosis
Acronym: TDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Castilla-La Mancha (Other)
Collaborators: Asociación Esclerosis Múltiple de Toledo, España (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GIFTO-ADEMTO
Record Dates: First submitted 2025-05-07; First posted 2025-05-22 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: tDCS; Sham tDCS
Keywords: tdcs; gait; multiple sclerosis; gait training
MeSH Terms: conditions — Multiple Sclerosis | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- tDCS (Experimental): Stimulation will be applied at an intensity of 2 mA for 20 minutes, with an average ramp-up and ramp-down rate of 0.1 mA/s, using circular electrodes of 35 cm² (resulting in a current density of 0.06 mA/cm²) covered with sponges moistened with 0.9% saline solution. A Sooma tDCS™ direct current stimulator (Sooma Oy Ltd, Helsinki, Finland), certified for clinical use, will be used. The anode will be placed over the Cz stimulation site, and the cathode will be placed on the right shoulder. The electrode will be secured to the participant's head using a neoprene cap (Neuroelectrics, Barcelona, Spain) and to the shoulder with a crepe bandage. Gait training will be performed using a treadmill and a body-weight support system consisting of a harness that also serves as a safety mechanism in case of a fall. Each session will last 20 minutes to allow for a sufficient number of gait cycles to promote motor relearning.
  Interventions: Device: tDCS
- Sham tDCS (Sham Comparator): The sham tDCS group will use the same device and electrode placement as the active stimulation group. The protocol will consist of a 10-second ramp-up to 1 mA, followed by a 7-second ramp-down to 0.3 mA, which will be maintained for 19 minutes and 40 seconds, and a final 3-second ramp-down to 0 mA. This sham stimulation method is integrated into the Sooma stimulator. Gait training will be performed using a treadmill and a body-weight support system consisting of a harness that also serves as a safety mechanism in case of a fall. Each session will last 20 minutes to allow for a sufficient number of gait cycles to promote motor relearning.
  Interventions: Device: shamtDCS

INTERVENTIONS:
Device: tDCS — Stimulation will be applied at an intensity of 2 mA for 20 minutes, with an average ramp-up and ramp-down rate of 0.1 mA/s, using rectangular electrodes of 35 cm² (resulting in a current density of 0.06 mA/cm²) covered with sponges moistened with 0.9% saline solution. A Sooma tDCS™ direct current stimulator (Sooma Oy Ltd, Helsinki, Finland), certified for clinical use, will be used. The anode will be placed over the Cz stimulation site, and the cathode will be placed on the right shoulder. The electrode will be secured to the participant's head using a neoprene cap (Neuroelectrics, Barcelona, Spain) and to the shoulder with a crepe bandage.
  Arms: tDCS
Device: shamtDCS — The sham tDCS group will use the same device and electrode placement as the active stimulation group. The protocol will consist of a 10-second ramp-up to 1 mA, followed by a 7-second ramp-down to 0.3 mA, which will be maintained for 19 minutes and 40 seconds, and a final 3-second ramp-down to 0 mA. This sham stimulation method is integrated into the Sooma stimulator.
  Arms: Sham tDCS

SUMMARY:
This clinical trial aims to evaluate the therapeutic effectiveness of transcranial direct current stimulation (tDCS), a non-invasive technique that modulates cortical excitability, in combination with gait training in patients with multiple sclerosis (MS). The study focuses on improving balance and walking ability, which are commonly impaired in this population. A randomized, triple-blind, controlled design will be used, comparing an active tDCS group with a sham stimulation group, both receiving the same gait training protocol. Outcomes will include functional and clinical measures related to mobility, balance, and fatigue. The project builds on previous meta-analytical evidence suggesting positive effects of tDCS in MS and aims to confirm these findings using an optimized stimulation protocol.

ELIGIBILITY:
Inclusion Criteria:

* Ability to understand and follow instructions.
* Diagnosis of Multiple Sclerosis according to McDonald criteria.
* Expanded Disability Status Scale (EDSS) between 1 and 6.
* Stable condition in the last three months.

Exclusion Criteria:

* Peripheral neurological injury of lower limbs.
* Metal objects in the head.
* Uncontrolled epilepsy.
* Diagnosis of psychiatric disorder.
* Fractures or fissures in the skull.
* Presence of any implanted electronic device (pacemaker, baclofen pump).
* Presence of ulcers in the harness attachment area.
* Osteoporotic fractures in the last 2 years.
* Height > 190 cm.
* Weight > 120 kg.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2025-05-26 (Estimated); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
TUG | Pre intervention, at the end of 10th session, and follow-up at 4 weeks
  Timed Up and Go (TUG) Test: Measures the time it takes for the patient to safely stand up from a chair with armrests, walk three meters to a marked line, turn around, return to the chair, and sit down. The patient may use assistive devices if needed.
Timed 25-Foot Walk | Pre intervention, at the end of 10th session, and follow-up at 4 weeks
  Timed 25-Foot Walk (T25-FW): Assesses gait speed by measuring the time it takes for a patient to walk a distance of 25 feet.

SECONDARY OUTCOMES:
MSWS-12 | Pre intervention, at the end of 10th session, and follow-up at 4 weeks
  12-Item Multiple Sclerosis Walking Scale (MSWS-12): A patient-reported outcome measure that assesses self-perceived walking ability by asking about mobility-related aspects over the past 15 days. Values: 12 up to 60. Higher scores mean worse walking ability.
FSS | Pre intervention, at the end of 10th session, and follow-up at 4 weeks
  Fatigue severity scale. The FSS measures the severity of fatigue and its impact on daily functioning. Scores range from 9 to 63, with higher scores reflecting more severe fatigue.

OTHER OUTCOMES:
Adverse events | 24 hours after the stimulation
  Questionnaire for adverse events
Borg | Before stimulation and just immediately after stimulation ends
  "Modified Borg Scale. It measures the perception of effort and the intensity of physical activity on a scale from 0 (complete rest) to 10 (maximum effort)."

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Asociación de Esclerosis Múltiple de Toledo, Toledo, Toledo
  - Universidad de Castilla La Mancha, Toledo, Toledo

IPD SHARING:
Plan to Share IPD: Yes
Scientific Journal